CLINICAL TRIAL: NCT05100836
Title: SURPASS Study - The Surgical Unloading Renal Protection And Sustainable Support Study
Brief Title: SURPASS Impella 5.5 Study
Status: Completed | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Surpass
Record Dates: First submitted 2021-10-12; First posted 2021-10-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cardiogenic Shock; Acute Decompensated Heart Failure
Keywords: Impella; Impella 5.5; Bridge to next therapy
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Single arm all comers supported with Impella 5.5
  Interventions: Device: Impella 5.5

INTERVENTIONS:
Device: Impella 5.5 — Impella 5.5 mechanical circulatory support

SUMMARY:
A multi-center, prospective & retrospective, observational single-arm study of the clinical outcomes up to one year collected from electronic health records of patients which have undergone standard of care implantation of Impella 5.5, regardless of clinical situation or indication. All patients will be enrolled via an IRB-approved Waiver of Informed Consent and HIPAA Authorization.

All patients who were supported retrospectively (prior to site IRB approval) with Impella 5.5 at the investigative site will be entered into the SURPASS registry and specified as the retrospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Subject has previously undergone an Impella 5.5 implant at a study site

Exclusion Criteria:

* Patients not receiving Impella 5.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and older who previously received an Impella 5.5 implant at the study site
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Survival Outcome | One year
  The rate of patients who survived at Impella 5.5 explant, hospital discharge and follow-up up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Funamoto, MD, Principal Investigator — Methodist San Antonio Hospital; Mark Anderson, MD, Principal Investigator — Hackensack Meridian Health; David D'Alessandro, MD, Principal Investigator — MGH; Gundars Katlaps, MD, Principal Investigator — Tampa General Hospital; Anthony Lemaire, MD, Principal Investigator — Robert Wood Johnson University Hospital; Edward Soltesz, MD, Principal Investigator — The Cleveland Clinic; Masashi Kawabori, MD, Principal Investigator — Tufts Medical Center; Ahmad Zeeshan, MD, Principal Investigator — Advent Health Orlando; Fardad Esmailian, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (15):
- United States (15):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Advent Health Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - MGH, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Integris Health Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist San Antonio Hospital, San Antonio, Texas